CLINICAL TRIAL: NCT02445794
Title: A Randomized, Double-blind, Controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of RT001 in Patients With Friedreich's Ataxia
Brief Title: A First in Human Study of RT001 in Patients With Friedreich's Ataxia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT001-002
Record Dates: First submitted 2015-05-06; First posted 2015-05-15 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-09

CONDITIONS: Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Cohort Studies; RT001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RT001, oral, 1.8 g/day (Experimental): RT001, oral, 1.8 g QD for 28 days or matching comparator
  Interventions: Drug: Low dose cohort; Drug: High dose cohort
- RT001, oral, 9 g/day (Experimental): RT001, oral, 4.5 g BID for 28 days or matching comparator
  Interventions: Drug: Low dose cohort; Drug: High dose cohort

INTERVENTIONS:
Drug: Low dose cohort — RT001 is encapsulated di-deutero synthetic homologue of linoleic acid ethyl ester. Each capsule contains 900 mg of RT001.
  Other Names: RT001 1.8 g/d (2 capsule per day); RT001 comparator 1.8 g/d (2 capsule per day)
Drug: High dose cohort — RT001 comparator is encapsulated non-deuterated linoleic acid ethyl ester.
  Other Names: RT001 9.0 g/d (9 capsule per day); RT001 comparator 9.0 g/d (9 capsule per day)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of RT001 in patients with Friedreich's ataxia.

DETAILED DESCRIPTION:
Study RT001-002 is a randomized, double-blind, controlled, ascending dose study to evaluate the safety, tolerability, pharmacokinetic, disease state, and exploratory endpoints in patients with Friedreich's ataxia after oral administration. The study includes 2 dose levels of RT001.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 50 years of age
2. Medical history consistent with the symptoms of FRDA at ≤ 25 years of age
3. Homozygous for GAA repeat expansions in the Frataxin gene in the affected range for FRDA
4. FARS-Neurological score of 20-90 points
5. Ambulatory (with or without assistive device) and capable of performing assessments/evaluations
6. Body Mass Index ≤ 29.9 kg/m2
7. Agrees to dietary restrictions and agrees to receive calls from a dietary coach
8. Signed the informed consent form prior to entry into the study
9. Agrees to spend the required number of overnight clinic days
10. Able to provide the necessary repeated blood samples

Exclusion Criteria:

1. Received treatment with other experimental therapies within the last 30 days prior to the first dose
2. Known point mutation in the FXN gene
3. History of malignancies (other than basal cell carcinomas)
4. Impaired renal function at screening
5. Alanine transaminase (ALT) or aspartate transaminase (AST) laboratory values > 2 x upper limit of normal (ULN) at screening
6. Known hepatitis B surface antigen (HBsAg)-positive, or known or suspected active hepatitis C infection, or is known to be human immunodeficiency virus (HIV) positive
7. Female who is breastfeeding or has a positive pregnancy test
8. Male participant or female participant of child bearing potential, who is sexually active and unwilling/unable to use a medically acceptable and effective double barrier birth control method throughout the study
9. Unwilling or unable to comply with the requirements of the protocol
10. Clinically significant cardiac abnormalities at screening that, in the opinion of the Investigator, would make the patient unsuitable for enrollment
11. Diabetes mellitus (Type 1 or 2)
12. Suicidal ideation as determined by the Columbia-Suicide Severity Rating Scale
13. History, within the last 2 years, of alcohol abuse, significant mental illness, or physical opioid dependence
14. Cannot adhere to the dietary guidance required to be followed by the protocol
15. Cannot take the medication due to impairment in swallowing capsules

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Scribner, MD, Study Director — Biojiva LLC; Theresa Zesiewicz, MD, Principal Investigator — USF Ataxia Research Center
Locations (2):
- United States (2):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - University of South Florida, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - RT001 (1.8 g/Day): RT001, oral, 2 capsules/day
  RT001: RT001 is encapsulated di-deutero synthetic homologue of linoleic acid ethyl ester. Each capsule contains 900 mg of RT001.
- Cohort 1 - Comparator: RT001 comparator, oral, 2 capsules/day
  RT001 comparator: RT001 comparator is encapsulated non-deuterated linoleic acid ethyl ester.
- Cohort 2 - RT001 (9 g/Day): RT001, oral, 10 capsules/day
  RT001: RT001 is encapsulated di-deutero synthetic homologue of linoleic acid ethyl ester. Each capsule contains 900 mg of RT001.
- Cohort 2 - Comparator: RT001 comparator, oral, 10 capsules/day
  RT001 comparator: RT001 comparator is encapsulated non-deuterated linoleic acid ethyl ester.
Period: Overall Study
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 1 - Comparator | Cohort 2 - RT001 (9 g/Day) | Cohort 2 - Comparator
Started | 6 | 3 | 7 | 3
Completed | 6 | 3 | 5 | 3
Not Completed | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - RT001: RT001 - 2 capsules/day (1.8 g/day)
- Cohort 1 - Comparator: RT001 comparator - 2 capsules/day
- Cohort 2 - RT001: RT001 - 10 capsules/day (9 g/day)
- Cohort 2 - Comparator: RT001 comparator - 10 capsules/day
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - RT001 | Cohort 1 - Comparator | Cohort 2 - RT001 | Cohort 2 - Comparator | Total
Number analyzed (Participants) | 6 | 3 | 7 | 3 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (7.61) | 45.3 (2.08) | 28.6 (7.46) | 26.3 (4.16) | 34.3 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 5 | 1 | 10
  Male | 3 | 2 | 2 | 2 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 3 | 7 | 3 | 19
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.82 (3.857) | 26.17 (2.798) | 21.63 (3.096) | 24.63 (7.931) | 23.47 (4.128)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 1 - Comparator | Cohort 2 - RT001 (9 g/Day) | Cohort 2 - Comparator
Number analyzed (Participants) | 6 | 3 | 7 | 3
participants | 5 | 2 | 5 | 2

2. Secondary Outcome: Pharmacokinetics - Area Under the Concentration-time Curve After a Single Dose
Description: AUC 0-24 hours post-dose (Hours -1.0 to -0.5 (pre-breakfast, pre-dose), 0.5 (± 5 min), 1 (± 5 min), 1.5 (± 5 min), 2 (± 10 min), 4 (± 10 min) (pre-lunch), 6 (± 10 min), 8 (± 10 min), 12 (± 10 min), and 16 (± 30 min) Day 2: 24 hours following dosing on Day 1 (± 30 min; pre-breakfast, pre-dose) was measured for the low and high dose cohorts after a single dose of RT001
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ug*h/mL
Groups:
- RT001, Oral, 1.8 g/Day: RT001, oral, 1.8 g QD for 28 days or matching comparator
  RT001: RT001 is encapsulated di-deutero synthetic homologue of linoleic acid ethyl ester. Each capsule contains 900 mg of RT001.
  RT001 comparator: RT001 comparator is encapsulated non-deuterated linoleic acid ethyl ester.
- RT001, Oral, 9 g/Day: RT001, oral, 4.5 g BID for 28 days or matching comparator
  RT001: RT001 is encapsulated di-deutero synthetic homologue of linoleic acid ethyl ester. Each capsule contains 900 mg of RT001.
  RT001 comparator: RT001 comparator is encapsulated non-deuterated linoleic acid ethyl ester.
Arm/Group | RT001, Oral, 1.8 g/Day | RT001, Oral, 9 g/Day
Number analyzed (Participants) | 6 | 7
ug*h/mL | 524 (86) | 915 (251)

3. Secondary Outcome: Pharmacokinetics - Maximum Observed Plasma Concentration After a Single Dose
Description: Plasma levels were measured for the following time points: Day 1: Hours -1.0 to -0.5 (pre-breakfast, pre-dose), 0.5 (± 5 min), 1 (± 5 min), 1.5 (± 5 min), 2 (± 10 min), 4 (± 10 min) (pre-lunch), 6 (± 10 min), 8 (± 10 min), 12 (± 10 min), and 16 (± 30 min) Day 2: 24 hours following dosing on Day 1 (± 30 min; pre-breakfast, pre-dose) PK curves were constructed from these data and CMax measured on the curves for the low and high dose cohorts
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 2 - RT001 (9 g/Day)
Number analyzed (Participants) | 6 | 7
ug/mL | 35.9 (9.8) | 58.6 (16)

4. Secondary Outcome: Pharmacokinetics - Time to Reach Maximum Plasma Concentration After a Single Dose
Description: TMax measured for the low and high dose cohorts
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 2 - RT001 (9 g/Day)
Number analyzed (Participants) | 6 | 7
h | 6.05 (0) | 8.0 (0)

5. Secondary Outcome: Pharmacokinetics - Maximum Observed Plasma Concentration After Final Dose on Day 28
Description: After 28 days of dosing, the final dose of RT001 was administered, and PK samples were obtained at the following timepoints (all timepoints refer to final dose on Day 28):
  Day 28: Hours -1.0 to -0.5 (pre-breakfast, pre-dose on Day 28), 0.5 (± 5 min), 1 (± 5 min), 1.5 (± 5 min), 2 (± 10 min), 4 (± 10 min) (pre-lunch), 6 (± 10 min), 8 (± 10 min), 12 (± 10 min), and 16 (± 30 min) Day 29: Hours 24 (± 30 min; pre-breakfast) and 32 (± 30 min) hours following final dose on Day 28 Day 30: 48 hours following final dose on Day 28 (± 30 min; pre-breakfast) Day 31: 72 hours following final dose on Day 28 (± 30 min; pre-breakfast) PK curves were constructed, and CMax at 28 days was determined from these curves
Time Frame: Day 28-Day 31 (3 days)
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 2 - RT001 (9 g/Day)
Number analyzed (Participants) | 6 | 5
ug/mL | 91 (44.6) | 359.9 (31.6)

6. Secondary Outcome: Pharmacokinetics - Terminal Half-life Estimation After Final Dose on Day 28
Description: After 28 days of dosing, the final dose of RT001 was administered, and PK samples were obtained at the following timepoints (all timepoints refer to final dose on Day 28):
  Day 28: Hours -1.0 to -0.5 (pre-breakfast, pre-dose on Day 28), 0.5 (± 5 min), 1 (± 5 min), 1.5 (± 5 min), 2 (± 10 min), 4 (± 10 min) (pre-lunch), 6 (± 10 min), 8 (± 10 min), 12 (± 10 min), and 16 (± 30 min) Day 29: Hours 24 (± 30 min; pre-breakfast) and 32 (± 30 min) hours following final dose on Day 28 Day 30: 48 hours following final dose on Day 28 (± 30 min; pre-breakfast) Day 31: 72 hours following final dose on Day 28 (± 30 min; pre-breakfast) PK curves were constructed, and T1/2 at 28 days was determined from these curves
Time Frame: Day 28-Day 31 (3 days)
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 2 - RT001 (9 g/Day)
Number analyzed (Participants) | 6 | 5
h | 42.3 (9.77) | 30.3 (18.3)

7. Secondary Outcome: Change From Baseline at 28 Days in the Timed 25 Foot Walk (T25FW)
Description: The T25FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk.
  T25FW was measured at baseline and at 28 days. These data were compared.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 1 - Comparator | Cohort 2 - RT001 (9 g/Day) | Cohort 2 - Comparator
Number analyzed (Participants) | 6 | 3 | 6 | 3
sec | .503 (3.7751) | -1.87 (1.1653) | -7.475 (28.6458) | .608 (2.4182)

8. Secondary Outcome: Change From Baseline at 28 Days in the Friedreich Ataxia Rating Scale (FARS) - Neurological Score (Minimum Score 0, Maximum Score 125, Lower is Better)
Description: The FARS-neurological rating scale specifically developed and validated for Friedreich's Ataxia. The FARS-Neurological included evaluations of the neurological signs that specifically reflect neural substrates affected in patients with FA. Based on a neurological examination bulbar (11 points), upper limb coordination (36 points), lower limb coordination (16 points), peripheral nervous system (26 points), and upright stability (36 points) functions were assessed for individual sub-scores (11, 36, 16, 26, and 36) with a maximum score of 125 (Friedreich's Ataxia Study Group, Subramony et al., 2005, Lynch et al., 2006). FARS-Neurologic examinations were conducted by a qualified physician or health professional trained in the use of the FARS format. A lower score is better. The minimum score is 0, the maximum score is 125.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale maximum 125
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 1 - Comparator | Cohort 2 - RT001 (9 g/Day) | Cohort 2 - Comparator
Number analyzed (Participants) | 6 | 3 | 7 | 3
units on a scale maximum 125 | -6.22 (2.796) | -6.47 (4.768) | -3.3 (2.080) | -2 (3.464)

9. Secondary Outcome: Change From Baseline at 28 Days in Peak Workload for the Treated Population vs. the Comparator Population
Description: Peak workload was measured using cardiopulmonary exercise testing at baseline and after 28 days of treatment. The results of treatment were compared to baseline examination.
Time Frame: 28 days
Population: Subjects unable to start or complete the test were excluded from analysis. Treatment and comparator cohorts were pooled to allow for statistical analysis.
Measure: Median (Full Range); unit: watts/kg
Groups:
- RT001: RT001, oral (pooled 1.8 g/d + 9.0 g/d)
  RT001: RT001 is encapsulated di-deutero synthetic homologue of linoleic acid ethyl ester. Each capsule contains 900 mg of RT001.
- Cohort 1 - Comparator: RT001 comparator, oral
  RT001 comparator: RT001 comparator is encapsulated non-deuterated linoleic acid ethyl ester.
Arm/Group | RT001 | Cohort 1 - Comparator
Number analyzed (Participants) | 10 | 6
watts/kg | .08 [-.1 to .34] | -.08 [-.3 to 0]
Statistical Analysis 1: Comparison: RT001 vs Cohort 1 - Comparator; Test type: Superiority; p = .008, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Cohort 1 - RT001 (1.8 g/Day) | Cohort 1 - Comparator | Cohort 2 - RT001 (9 g/Day) | Cohort 2 - Comparator
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 1/7 | 0/3
Other Adverse Events (participants affected / at risk) | 5/6 | 2/3 | 5/7 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - RT001 (1.8 g/Day) (N=6) | Cohort 1 - Comparator (N=3) | Cohort 2 - RT001 (9 g/Day) (N=7) | Cohort 2 - Comparator (N=3)
Steatorrhea requiring overnight hospitalization (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 — The subject developed severe steatorrhea after a single dose of RT001. This required overnight hospitalization. The condition resolved after within 24 hours after drug discontinuation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - RT001 (1.8 g/Day) (N=6) | Cohort 1 - Comparator (N=3) | Cohort 2 - RT001 (9 g/Day) (N=7) | Cohort 2 - Comparator (N=3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Most of the TEAEs were mild gastrointestinal distress due to the fat content of the study drug (both active and the comparator.) They were self-limited.
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
facial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No